CLINICAL TRIAL: NCT02267239
Title: Methodology of Application and Immediate Effect of the Essential Oils and 0.2% Chlorhexidine on Oral Biofilm: Immersion Versus Mouthwash.
Brief Title: Methodology Antiseptic Application, Influence on Oral Biofilm.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior lecturer, University of Santiago de Compostela
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: immersion vs. mouthwash
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Oral Biofilm; Periodontitis; Gingivitis
Keywords: essential oils; chlorhexidine; microscopy, confocal; immersion; antiseptic
MeSH Terms: conditions — Periodontitis; Gingivitis | interventions — Oils, Volatile; Immersion; Listerine; Chlorhexidine; Mouthwashes; Tooth Exfoliation; Casts, Surgical; Models, Biological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Essential Oils, immersion (Active Comparator): Professional oral cleaning Plaster cast IDODS Immersion the disk with the biofilm in the essential oils antiseptic solution
  Interventions: Drug: essential oils, immersion; Procedure: professional oral cleaning; Procedure: Plaster cast; Device: IDODS
- Chlorhexidine, immersion (Active Comparator): Professional oral cleaning Plaster cast IDODS Immersion the disk with the biofilm in the chlorhexidine antiseptic solution
  Interventions: Drug: Chlorhexidine, immersion; Procedure: professional oral cleaning; Procedure: Plaster cast; Device: IDODS
- baseline (Other): Professional oral cleaning Plaster cast IDODS Disk in basal conditions.
  Interventions: Procedure: professional oral cleaning; Procedure: Plaster cast; Device: IDODS
- Essential Oils, mouthwash (Active Comparator): Professional oral cleaning Plaster cast IDODS Active mouthwash with the essential oils antiseptic solution
  Interventions: Drug: essential oils, mouthwash; Procedure: professional oral cleaning; Procedure: Plaster cast; Device: IDODS
- Chlorhexidine, mouthwash (Active Comparator): Professional oral cleaning Plaster cast IDODS Active mouthwash with the chlorhexidine antiseptic solution
  Interventions: Drug: chlorhexidine, mouthwash; Procedure: professional oral cleaning; Procedure: Plaster cast; Device: IDODS

INTERVENTIONS:
Drug: essential oils, immersion — A single, 30-second immersion in 1 mL of essential oils in a hydroalcoholic solution (Listerine Mentol, Listerine®, Johnson & Johnson, Madrid, Spain) (I-EO).
  Other Names: Listerine, Listerine Mentol, essential oil
  Arms: Essential Oils, immersion
Drug: Chlorhexidine, immersion — A single, 30-second immersion in 1 mL of 0.2% chlorhexidine (Oraldine Perio®, Johnson and Johnson, Madrid, Spain) (I-0.2% CHX).
  Other Names: Oraldine Perio
  Arms: Chlorhexidine, immersion
Drug: essential oils, mouthwash — A single, 30-second mouthwash with 20 mL of essential oils in a hydroalcoholic solution (Listerine Mentol, Listerine®, Johnson & Johnson, Madrid, Spain) (M-EO).
  Other Names: Listerine, Listerine Mentol, essential oil
  Arms: Essential Oils, mouthwash
Drug: chlorhexidine, mouthwash — A single, 30-second mouthwash with 10 mL of 0.2% chlorhexidine (Oraldine Perio®, Johnson and Johnson, Madrid, Spain) (M-0.2% CHX).
  Other Names: Oraldine perio
  Arms: Chlorhexidine, mouthwash
Procedure: professional oral cleaning — scaling and polishing teeth of the volunteers
  Other Names: tartrectomy, scaling and polishing
Procedure: Plaster cast — Taking a plaster cast of the volunteers' mouth
  Other Names: model, dental impresionss
Device: IDODS — Specific intraoral device which carries six glass disks
  Other Names: Intraoral Device of Overlaid Disk-holding Splints

SUMMARY:
The study has the objective to compare two different methodology of application the antiseptic on the oral biofilm will be formed during 48h in situ on a specific device. The first one using the immersion in the antiseptic solution, as much of the authors did in the past. And the second way doing a active mouthwash, as the manufacturer recommends.

The study will compare two different antiseptic solutions, the chlorhexidine (0.2% Oraldine Perio) and the essential oils (Listerine Mentol) with the two different application and compared the bacterial vitality, thickness and covering grade between solutions and with a basal sample.

DETAILED DESCRIPTION:
15 healthy volunteers, between 20 and 45 years old, will use during 48 hours two specific oral devices with 3 glass disks each. After this period, one of the disk will be drawn from the device and it will be immersed in Live/Dead BacLight solution for 15 minutes and then the disk will be analysed by the Confocal Laser Scanning Microscope (CLSM). Immediately, another disk will be removed from the intraoral device and immersed in the antiseptic solution, being analysed by the CLSM as well. After that, the volunteers will do the mouthwash with the antiseptic solution (as stated in the specific protocol) and the last disk will be drawn from the device and will be analysed by the CLSM following the same protocol. The other 3 disk will undergo the same protocol of baseline, immersion and mouthwash, but with the other antiseptic solution.

The CLSM data will be analysed and the bacterial vitality, thickness and covering grade will be calculated. Finally the statistical analysis will be applied (Pairwise comparisons, with the Bonferroni adjustment).

ELIGIBILITY:
Inclusion Criteria:

* good oral health status: a minimum of 24 permanent teeth with no evidence of gingivitis or periodontitis and absence of untreated caries

Exclusion Criteria:

* smoker or former smoker
* presence of dental prostheses or orthodontic devices
* antibiotic treatment or routine use of oral antiseptics in the previous three months
* presence of any systemic disease that could alter the production or composition of saliva

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
change in bacterial vitality | baseline, 30seconds after immersion and 30 seconds after mouthwash (in both antiseptic solutions)
  percentage of live bacteria in the sample
change in thickness | baseline, 30 seconds after immersion and 30 seconds after mouthwash (in both antiseptic solutions)
  maximum numbers of layers (1micra per layer) with continuous presence of bacteria
change in covering grade | baseline, 30seconds after immersion and 30 seconds after mouthwash (in both antiseptic solutions)
  percentage of the disk surface occupied by the biofilm

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Inmaculada, Senior lecturer, Study Director — Faculty of Medicine and Dentistry of the University of Santiago de Compostela Santiago de Compostela, A Coruña, Spain, 15782
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Derived] Prada-Lopez I, Quintas V, Casares-De-Cal MA, Suarez-Quintanilla JA, Suarez-Quintanilla D, Tomas I. Ex vivo vs. in vivo antibacterial activity of two antiseptics on oral biofilm. Front Microbiol. 2015 Jul 2;6:655. doi: 10.3389/fmicb.2015.00655. eCollection 2015. PMID 26191050